CLINICAL TRIAL: NCT02243735
Title: Multicenter Randomized Controlled Trial Comparing Ferric(III)Carboxymaltose Infusion With Oral Iron Suppletion in the Treatment of Preoperative Anaemia in Colorectal Cancer Patients
Brief Title: Trial Comparing Ferric(III)Carboxymaltose Infusion With Oral Iron Suppletion as Treatment of Anaemia
Acronym: FIT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Vifor Pharma (Industry)
Responsible Party: Principal Investigator, Prof. dr. W.A. Bemelman, Professor, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL50013.018.14; 2014-002827-87 (EudraCT Number)
Record Dates: First submitted 2014-09-12; First posted 2014-09-18 (Estimated); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Anemia; Colorectal Carcinoma; Surgery
MeSH Terms: conditions — Anemia; Colorectal Neoplasms | interventions — ferrous fumarate; ferric carboxymaltose

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ferrous fumarate (Active Comparator): Patients randomized to standard care with ferrous fumarate will receive three tablets of 200 mg daily from randomisation until day before surgery
  Interventions: Drug: Ferrous fumarate
- ferric(III)carboxymaltose (Active Comparator): Patients randomized to intravenous iron (ferric(III)carboxymaltose) will be dosed according to Summary of Product Characteristics (SPC) depending on body weight and Hb value and administered in one or two infusions with one week in between. A maximum dose of 1000mg or 15mg/kg per week will be administered
  Interventions: Drug: ferric(III)carboxymaltose

INTERVENTIONS:
Drug: Ferrous fumarate — Patients randomized to standard care with ferrous fumarate will receive three tablets of 200 mg daily from randomisation until day before surgery
  Other Names: ferrofumarate
  Arms: Ferrous fumarate
Drug: ferric(III)carboxymaltose — Patients randomized to intravenous iron (ferric(III)carboxymaltose) will be dosed according to Summary of Product Characteristics (SPC) depending on body weight and Hb value and administered in one or two infusions with one week in between. A maximum dose of 1000mg or 15mg/kg per week will be administered
  Other Names: Ferinject
  Arms: ferric(III)carboxymaltose

SUMMARY:
The aim of this multicenter trial is to determine the efficacy of preoperative intravenous iron suppletion in comparison with the standard preoperative oral substitution in anaemic patients with colorectal cancer in curing the anemia and the assess the effect of preoperative iron on morbidity, postoperative recovery and quality of life.

Hypothesis: It is our hypothesis that a more profound approach of preoperative anaemia with intravenous iron will lead to a higher percentage of patients with normalization of Hb-level (> 12 g/dl (7.5 mmol/l) for women and > 13 g/dl (8 mmol/l) for men), which potentially reduces morbidity, length of stay, improves quality of live, decreases fatigue and could be more cost effective compared to current practice with oral substitution of iron.

DETAILED DESCRIPTION:
This multicenter randomized clinical trial aims to optimize postoperative outcome in anaemic patients who undergo curative surgery for colorectal carcinoma. The aim of this trial is to investigate which route of administration is superior in the treatment of iron deficiency anaemia in these patients. In addition, an economic evaluation of intravenous iron versus oral iron will be done. The evaluation will be performed from a societal perspective as (i) a cost-effectiveness analysis with the costs per responder to iron suppletion therapy as primary outcome and (ii) a cost-utility analysis with the costs per quality adjusted life-year (QALY) as primary outcome. The cost effectiveness analysis closely relates to clinical efficacy measure and allows for setting priorities in treatment of anaemia in colorectal cancer patients. The cost-utility analysis allows for a comparison of the societal impact of intravenous iron suppletion on post-operative recovery, such as shorter length of stay and earlier return to daily activities, with the impact of other interventions and of interventions in other areas of health care.

The primary aim of this trial is:

1. To compare the percentage of patients with normalization of Hb-level (> 12 g/dl (7.5 mmol/l) for women and > 13 g/dl (8 mmol/l) for men after intravenous versus oral iron therapy in patients undergoing curative surgery for colorectal carcinoma.

   Secondary aims of the FIT trial are:
2. To analyse the effect of preoperative iron therapy (intravenous versus oral) on postoperative morbidity, length of stay, amount of blood transfusions needed and quality of life and fatigue scores.
3. To determine the cost effectiveness of preoperative intravenous iron substitution in comparison with oral substitution.

Sample size:

The principal analysis will consist of an intention-to-treat comparison of the proportions of patients with iron deficiency anaemia between the two study groups. The trial is designed as a superiority trial, hypothesizing a greater percentage of patients achieving normalization of Hb-level (called 'responder') in favour of infusion of ferric(III)carboxymaltose compared to oral iron suppletion. Our power calculation is based on the study of Seid et al(19), which compared ferric(III)carboxymaltose with oral ferrous sulphate in a population of post-partum women with an iron deficiency anaemia. The proportion achieving a normalization of Hb after two weeks of treatment was 55% in the intravenous iron group and 35% in the oral iron group. We expect that the efficacy of the iron therapy is lower in patients with a colorectal carcinoma. Therefore, the expected percentage of patients who achieve normalization of Hb-level (Hb >7.5 mmol/l (12 g/dl) for women and Hb >8.o mmol/l (13 g/dl) for men) is 45% in the intravenous iron group and 25% in the oral iron group. Based on these proportions, a sample size of 89 patients per group is needed for a Chi square test to achieve 80% power at a two sided alpha of 0.05. With an estimated loss to follow up of 10%, a sample size of 198 is calculated. We used nQuery advisor version 7.0 to calculate the sample size.

ELIGIBILITY:
Inclusion Criteria:

* M0-stage Colorectal carcinoma
* Laparoscopic or open segmental colonic resection or (low) anterior resection
* Iron deficiency anaemia: Hb <7,5 mmol/l (12 g/dl) for women and Hb < 8 mmol/l (13 g/dl) for men and TSAT<20%
* Age 18 or older
* Written informed consent for study participation

Exclusion Criteria:

* Palliative surgery / metastasized disease
* Received blood transfusion within one month before screening
* Serum ferritin ≥ 800 µg/L
* Pregnancy
* Preoperative chemoradiation (Short course radiotherapy (5x5 Gy) = no exclusion)
* Contraindication for the use of ferric(III)carboxymaltose or ferrofumarate
* ASA classification > 3
* Use of erythropoietin stimulating agents within three months before screening
* Chronic kidney disease (GFR < 30ml/min/m)
* Myelodysplastic syndrome
* Severe anaemia with indication for blood transfusion
* Elevated liver enzymes (more than three times normal value)
* Hereditary Hemochromatosis
* Thalassemia
* Haemolytic anaemia/ chronic haemolysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2014-11; Primary Completion 2019-11 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Normalization of Hb-level. | From Baseline (date of randomisation) untill day of admission for surgery
  Percentage of patients with normalization of Hb-level from start treatment until day of admission for surgery. (Hb >12g/dl (7.5mmol/L) for women and Hb >13 g/dl (8.0mmol/L) for men).
  Patient will be randomised after they visit the surgery outpatient clinic to discuss the treatment option for their colorectal carcinoma. Average time between this visit and surgery in the Netherlands is maximally 5 weeks. Patients on oral iron suppletion will start with the iron therapy on the day of the randomisation. For the patients that will receive intravenous iron an appointment will be made on the short-care unit to facilitate the infusion of the iron. The period between infusion and surgery should be longer than two weeks.
  Our primary endpoint: Percentage of patients with normalization of Hb-level. Will be measured at the day of admission before surgery. Which is one day prior to surgery. The Hb-level will be followed-up after surgery on postoperative day 1, day 7 and after 4,8 and 12 weeks.

SECONDARY OUTCOMES:
Difference in Morbidity score | postoperative at week 1, week 4, week 8 and week 12
  The difference in morbidity score will be assessed using the Comprehensive Complication index, between both study groups

CONTACTS AND LOCATIONS:
Overall Officials: W. A Bemelman, Proffessor, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (13):
- Netherlands (13):
  - Medisch Centrum Alkmaar, Alkmaar
  - Flevoziekenhuis, Almere Stad
  - Meander Ziekenhuis, Amersfoort
  - Academic Medical Center, Amsterdam
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Sint Lucas Andreas Ziekenhuis, Amsterdam
  - Spaarne ziekenhuis, Amsterdam
  - VU medical center, Amsterdam
  - Amsterdam
  - Gelre Ziekenhuis, Apeldoorn
  - Albert Schweizer Ziekenhuis, Dordrecht
  - Tergooi ziekenhuis, Hilversum
  - Haga Ziekenhuis, The Hague

REFERENCES:
- [Derived] Talboom K, Borstlap WAA, Roodbeen SX, Bruns ERJ, Buskens CJ, Hompes R, Tytgat KMAJ, Tuynman JB, Consten ECJ, Heuff G, Kuiper T, van Geloven AAW, Veldhuis GJ, van der Hoeven JAB, Gerhards MF, Sietses C, Spinelli A, van de Ven AWH, van der Zaag ES, Westerterp M, van Westreenen HL, Dijkgraaf ML, Juffermans NP, Bemelman WA; FIT collaborative group. Ferric carboxymaltose infusion versus oral iron supplementation for preoperative iron deficiency anaemia in patients with colorectal cancer (FIT): a multicentre, open-label, randomised, controlled trial. Lancet Haematol. 2023 Apr;10(4):e250-e260. doi: 10.1016/S2352-3026(22)00402-1. Epub 2023 Feb 27. PMID 36863386
- [Derived] Borstlap WAA, Buskens CJ, Tytgat KMAJ, Tuynman JB, Consten ECJ, Tolboom RC, Heuff G, van Geloven N, van Wagensveld BA, C A Wientjes CA, Gerhards MF, de Castro SMM, Jansen J, van der Ven AWH, van der Zaag E, Omloo JM, van Westreenen HL, Winter DC, Kennelly RP, Dijkgraaf MGW, Tanis PJ, Bemelman WA. Multicentre randomized controlled trial comparing ferric(III)carboxymaltose infusion with oral iron supplementation in the treatment of preoperative anaemia in colorectal cancer patients. BMC Surg. 2015 Jun 28;15:78. doi: 10.1186/s12893-015-0065-6. PMID 26123286